CLINICAL TRIAL: NCT02094898
Title: Acute and Maintenance Intravenous Ketamine for Treatment Resistant Major Depression With Suicidal Ideation/Attempt
Brief Title: Ketamine for Depression and Suicide Risk
Acronym: Ketamine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William V. Bobo, M.D., Consultant - Psychiatry, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-005152
Record Dates: First submitted 2014-03-10; First posted 2014-03-24 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Depression; Suicide
Keywords: Depression; Unipolar; Bipolar; Suicidal
MeSH Terms: conditions — Depression; Suicide | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine infusion (Experimental): This trial was conducted in 2 phases. During the acute-phase, i.v. ketamine was administered thrice-weekly for up to 2 weeks.Those who achieved depressive symptom remission received continuation-phase treatment that consisted of once-weekly i.v. ketamine infusions for 4 additional weeks. Remission could occur after any of the 6 acute-phase infusions, at which point the next infusion was the first (of four) continuation-phase infusions. Individuals who remitted during acute-phase and completed continuation-phase treatment had 4 additional weekly post-continuation follow-up visits.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 0.3 mg/kg/hr of ketamine infused for 100 minutes
  Other Names: Ketalar

SUMMARY:
The purpose of this research study was to find out if the medication known as ketamine could help the symptoms of depression. This drug is approved by the U.S. Food and Drug Administration (FDA) as an anesthetic agent; however, it is not approved for use in depression treatment. The FDA allowed the use of this drug in this research study.

DETAILED DESCRIPTION:
This was a single-arm, open-label trial conducted in two phases. During the acute-phase, i.v. ketamine was administered thrice-weekly for up to 2 weeks.Those who achieved depressive symptom remission (Montgomery Åsberg Depression Rating Scale (MÅDRS)) total score less than or equal to 9 measured 24h after any acute-phase infusion) received continuation-phase treatment that consisted of once-weekly i.v. ketamine infusions for 4 additional weeks. Remission could occur after any of the 6 acute-phase infusions, at which point the next infusion was the first (of four) continuation-phase infusions. Individuals who remitted during acute-phase and completed continuation-phase treatment had 4 additional weekly post-continuation follow-up visits.Those who responded to i.v. ketamine (less than or equal to 50% reduction from baseline in MÅDRS total score) but did not remit during acute-phase were not eligible for continuation-phase treatment. Suicidal ideation was assessed clinically throughout the trial, supplemented by scores on the MÅDRS suicide item.

ELIGIBILITY:
Inclusion Criteria:

* Current psychiatric hospital inpatient at Mayo Clinic at time of initiation of treatment.
* Ability to provide informed consent
* Male/Female
* Age 18-65 yrs.
* Major Depressive Disorder or Bipolar Disorder I or Bipolar Disorder II with Patient Health Questionnaire-9 (PHQ 9) score ≥15 at hospital assessment
* Treatment resistant depression (TRD) as defined by at least two previous antidepressant or mood stabilizing treatments for depression in adequate dose for 8 weeks
* Patient reported overall suicide risk score ≥3 on the Suicide Status Form (SSF II-R) or score of ≥1on Item 9 of PHQ-9 (all at admission assessment)
* Ability to pass comprehension assessment test related to effects of ketamine and trial objectives and criteria
* Voluntary admission

Exclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, or active psychosis
* Index episode of depression greater than 2 years
* Ongoing prescription of ≥4 mg lorazepam equivalents total daily or a.m. dosing of any benzodiazepine at time of assessment
* Currently undergoing electroconvulsive therapy, deep brain stimulation or transcranial magnetic stimulation as acute series or for maintenance
* Any active or unstable medical condition as judged by principal investigator
* Previous use or abuse of methamphetamine, cocaine, stimulants (prescribed and illicit) within past 12 months
* Any current abuse or dependence of alcohol or drugs (except nicotine) and abuse or dependence of drugs and alcohol only in full remission (> 1 month, < 12 months). Patients will be allowed to enroll if their drug and alcohol abuse / dependence is in full (complete, not partial) sustained (> 1 year) remission.
* History of traumatic brain injury
* Developmental delay and intellectual disorder
* Encephalopathy (clinical diagnosis within prior 12 months of delirium)
* Cognitive disorder (mild and major)
* Previous participation in earlier Ketamine trial
* Pregnancy
* Prisoners
* Involuntarily hospitalized

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William V Bobo, MD, Principal Investigator — Consultant - Psychiatry
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vande Voort JL, Morgan RJ, Kung S, Rasmussen KG, Rico J, Palmer BA, Schak KM, Tye SJ, Ritter MJ, Frye MA, Bobo WV. Continuation phase intravenous ketamine in adults with treatment-resistant depression. J Affect Disord. 2016 Dec;206:300-304. doi: 10.1016/j.jad.2016.09.008. Epub 2016 Sep 12. PMID 27656788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Mayo Clinic in Rochester, Minnesota between 12/30/14 and 5/18/16.
Period: Overall Study
Arm/Group | Ketamine Infusion
Started | 12
Completed | 7
Not Completed | 5
Not completed — Clinical Worsening | 2
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine Infusion
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: MADRS Total Score at Baseline and Last Acute Phase Observation
Description: The Montgomery Asberg Depression Scale (MADRS) is a 10-item observer rating scale assessing symptoms of depression. The score ranges from 0 (no depression) to 60 (very depressed). For this study a score of less than or equal to 9 was considered clinical remission of depression.
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Entire Cohort: All enrolled subjects receiving at least one acute-phase ketamine infusion.
- Remission: Remission was defined as a MADRS total score of less than or equal to 9 measured 24 hours after any acute phase infusion.
- Non-Remission: Subjects who did not have a MADRS total score less than or equal to 9 measured 24 h after any acute phase infusion
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
units on a scale
  Baseline | 29.4 (7.5) | 29.4 (8.2) | 29.4 (7.7)
  Last acute phase observation | 15.9 (10.6) | 5.4 (3.4) | 23.4 (6.3)
Statistical Analysis 1: Comparison: Entire Cohort; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.05, t-test, 2 sided

2. Secondary Outcome: MADRS Total Score, Percent Change From Baseline at Last Acute Phase Observation
Description: as for outcome 1
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: percentage change in score
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
percentage change in score | -41.5 (40.3) | -79.1 (13.0) | -14.5 (11.0)
Statistical Analysis 1: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.001, t-test, 2 sided

3. Secondary Outcome: MADRS Factor 1 Score at Baseline and Last Acute Phase Observation
Description: The MADRS test includes 10 items and uses a 0 to 6 severity scale for each item, with higher scores indicating increasing depressive symptoms. MADRS Factor 1 (Sadness) consisted of MADRS items 1 (Apparent Sadness) and 2 (Reported Sadness). The MADRS Factor 1 Score is derived by adding all the scores from the 2 items, meaning the lowest possible score is 0 and the highest possible is 12.
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
units on a scale
  Baseline | 7.4 (2.0) | 7.4 (2.6) | 7.4 (1.7)
  Last acute phase observation | 3.5 (2.3) | 1.2 (0.5) | 5.1 (0.5)
Statistical Analysis 1: Comparison: Entire Cohort; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: Non-Remission; alpha level of 0.05; Test type: Superiority; p < 0.08, t-test, 2 sided

4. Secondary Outcome: MADRS Factor 1 Score, Percent Change From Baseline at Last Acute Phase Observation
Description: as for outcome 3
Time Frame: baseline, last acute phase observation
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: percentage change in score
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
percentage change in score | -50.3 (35.7) | -83.6 (15.7) | -26.5 (24.2)
Statistical Analysis 1: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.001, t-test, 2 sided

5. Secondary Outcome: MADRS Factor 2 Score at Baseline and Last Acute Phase Observation
Description: The MADRS test includes 10 items and uses a 0 to 6 severity scale for each item, with higher scores indicating increasing depressive symptoms. MADRS Factor 2 (Negative Thoughts) consisted of MADRS items 9 (Pessimistic Thoughts) and 10 (Suicidal Thoughts). The MADRS Factor 2 Score is derived by adding all the scores from the 2 items, meaning the lowest possible score is 0 and the highest possible is 12.
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
units on a scale
  Baseline | 6.0 (1.5) | 6.2 (1.6) | 5.9 (1.6)
  Last acute phase observation | 3.4 (1.7) | 1.8 (1.5) | 4.6 (0.5)
Statistical Analysis 1: Comparison: Entire Cohort; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.08, t-test, 2 sided

6. Secondary Outcome: MADRS Factor 2 Score, Percentage Change From Baseline at Last Acute Phase Observation
Description: as for outcome 5
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: percentage change in score
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
percentage change in score | -37.0 (36.5) | -65.4 (31.4) | -16.7 (25.2)
Statistical Analysis 1: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided

7. Secondary Outcome: MADRS Factor 3 Score at Baseline and Last Acute Phase Observation
Description: The MADRS test includes 10 items and uses a 0 to 6 severity scale for each item, with higher scores indicating increasing depressive symptoms. MADRS Factor 3 (Detachment) consisted of MADRS items 6 - 8 (Concentration Difficulties, Lassitude, and Inability to Feel). The MADRS Factor 3 Score is derived by adding all the scores from the 3 items, meaning the lowest possible score is 0 and the highest possible is 18.
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
units on a scale
  Baseline | 9.5 (3.1) | 9.8 (2.7) | 9.3 (3.5)
  Last acute phase observation | 4.9 (3.5) | 1.4 (1.3) | 7.4 (1.8)
Statistical Analysis 1: Comparison: Entire Cohort; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided

8. Secondary Outcome: MADRS Factor 3 Score, Percentage Change From Baseline at Last Acute Phase Observation
Description: as for outcome 7
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: percentage change in score
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
percentage change in score | -40.2 (48.5) | -84.3 (14.8) | -8.9 (37.3)
Statistical Analysis 1: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided

9. Secondary Outcome: MADRS Factor 4 Score at Baseline and Last Acute Phase Observation
Description: The MADRS test includes 10 items and uses a 0 to 6 severity scale for each item, with higher scores indicating increasing depressive symptoms. MADRS Factor 4 (Neurovegetative Symptoms) consisted of MADRS items 3-5 (Inner Tension, Reduced Sleep, and Reduced Appetite). The MADRS Factor 4 Score is derived by adding all the scores from the 3 items, meaning the lowest possible score is 0 and the highest possible is 18.
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
units on a scale
  Baseline | 6.5 (3.0) | 6.0 (3.8) | 6.9 (2.6)
  Last acute phase observation | 3.8 (3.6) | 1.0 (1.2) | 5.9 (3.4)
Statistical Analysis 1: Comparison: Entire Cohort; alpha level of 0.05; Test type: Superiority; p < 0.08, t-test, 2 sided
Statistical Analysis 2: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.08, t-test, 2 sided

10. Secondary Outcome: MADRS Factor 4 Score, Percentage Change From Baseline at Last Acute Phase Observation
Description: as for outcome 9
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: percentage change in score
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
percentage change in score | -36.0 (58.0) | -84.3 (20.4) | -8.4 (54.4)
Statistical Analysis 1: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.001, t-test, 2 sided

11. Secondary Outcome: MADRS Suicide Thoughts (Item 10) Score at Last Acute Phase Observation
Description: The MADRS test includes 10 items and uses a 0 to 6 severity scale for each item, with higher scores indicating increasing depressive symptoms. Item 10 scores can range from 0 to 6 (with 0 indicating enjoying life, and 6 indicating explicit plans for suicide.)
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
units on a scale
  Baseline | 2.9 (1.1) | 3.2 (1.1) | 2.7 (1.1)
  Last acute phase observation | 1.7 (0.8) | 1.2 (0.8) | 2.2 (0.4)
Statistical Analysis 1: Comparison: Entire Cohort; alpha level of 0.05; Test type: Superiority; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.08, t-test, 2 sided

12. Secondary Outcome: MADRS Suicide (Item 10) Score, Percentage Change From Baseline at Last Acute Phase Observation
Description: as for outcome 11
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: percentage change in score
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
percentage change in score | -26.7 (45.4) | -50.0 (46.8) | -7.2 (37.1)
Statistical Analysis 1: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.001, t-test, 2 sided

13. Secondary Outcome: Clinical Global Impression-severity Subscale (CGI-S) at Baseline and Last Acute Phase Observation
Description: The Clinical Global Impression Severity Subscale is an observer rated scale that measures illness severity. It has a range of responses from 1 (normal) through to 7 (among the most extremely ill patients).
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
units on a scale
  Baseline | 5.6 (0.5) | 5.4 (0.5) | 5.7 (0.5)
  Last acute phase observation | 3.9 (1.7) | 2.6 (0.9) | 4.9 (1.6)
Statistical Analysis 1: Comparison: Entire Cohort; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Remission; alpha level of 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided

14. Secondary Outcome: CGI-S Score, Percentage Change From Baseline at Last Acute Phase Observation
Description: as for outcome 13
Time Frame: baseline, last acute phase observation (approximately 2 weeks)
Population: Statistical analyses included all subjects who received at least one acute-phase ketamine infusion.
Measure: Mean (Standard Deviation); unit: percentage change in score
Arm/Group | Entire Cohort | Remission | Non-Remission
Number analyzed (Participants) | 12 | 5 | 7
percentage change in score | -29.4 (30.8) | -50.7 (20.3) | -14.3 (28.7)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Ketamine Infusion
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Infusion (N=12)
Clinical worsening - behavioral outburst and suicide threats (Psychiatric disorders) | 1 (1)
Suicide (Psychiatric disorders) | 1 (1) — Subject died by suicide 10 weeks after being withdrawn from the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Infusion (N=12)
Dissociation (Psychiatric disorders) | 9 (9)
Dizziness (General disorders) | 7 (7)
Numbness or tingling in extremities (General disorders) | 7 (7)
Sleepiness or sedation (General disorders) | 6 (6)
tearfulness/emotionality (Psychiatric disorders) | 4 (4)
Facial numbness (Nervous system disorders) | 3 (3)
Transient increases in systolic blood pressure (Blood and lymphatic system disorders) | 12 (12)
Transient increases in diastolic blood pressue (Blood and lymphatic system disorders) | 12 (12)

LIMITATIONS AND CAVEATS:
Lack of placebo or other control group and small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes